CLINICAL TRIAL: NCT04851340
Title: Validation of a Proprietary Test Strip for the Detection of Bovine and Soy Proteins in Human Milk: a Randomized Crossover Study
Brief Title: Investigating the Detection of Bovine and Soy Proteins in Human Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: Free to Feed Inc. (Unknown)
Responsible Party: Principal Investigator, Michelle McGuire, Director of Margaret Ritchie School of Family and Consumer Sciences, University of Idaho
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-126
Record Dates: First submitted 2020-12-01; First posted 2021-04-20 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2022-03

CONDITIONS: Microbiome; Stress; Food Allergy in Infants
Keywords: Food Allergy; Breastfeeding; Maternal Stress; Microbiome
MeSH Terms: conditions — Food Hypersensitivity; Breast Feeding | interventions — Milk; Soy Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cow's Milk First (Experimental): Participants in this group will eliminate all cow's milk products during the first 10 days of the study and receive the cow's milk intervention first and then will cross-over to eliminate soy products in the second 10 days of the study and receive the soy milk intervention during the second diet intervention.
  Interventions: Other: Cow's Milk; Other: Soy Milk
- Soy Milk First (Experimental): Participants in this group will eliminate all soy products during the first 10 days of the study and receive the soy milk intervention first and then will cross-over to eliminate cow's milk products in the second 10 days of the study and receive the cow's milk intervention during the second diet intervention.
  Interventions: Other: Cow's Milk; Other: Soy Milk

INTERVENTIONS:
Other: Cow's Milk — Participants will consume 200 mL, 300 mL, and 400 mL of 1% bovine milk during the diet challenge which occurs on three consecutive days of the study. The first day of the diet challenge participants consume 200 mL, the second day 300 mL and the third day 400 mL.
Other: Soy Milk — Participants will consume 200 mL, 300 mL, and 400 mL of soy milk during the diet challenge which occurs on three consecutive days of the study. The first day of the diet challenge participants consume 200 mL, the second day 300 mL and the third day 400 mL.

SUMMARY:
This study is a randomized, cross-over, dietary intervention research design comprising a 5-day run-in period, two 3-day dietary interventions, and a 2-day washout period. Participants (mother-offspring dyads) will be randomly assigned to order of interventions. Participants will be recruited as a convenience sample from mother-offspring dyads in the greater Moscow, Idaho and Boise, Idaho areas. The initial purpose of this study is to to learn more about the use of an allergen test strip to detect cow's milk and soy food allergen proteins in human milk, to identify soy and bovine-derived peptides in human milk after consumption of these foods, to explore the impact of maternal bovine milk and soy milk consumption on human milk and maternal/infant gastrointestinal microbiomes and to examine maternal stress during periods of dietary elimination and re-introductions periods.

DETAILED DESCRIPTION:
The current estimated prevalence of Immunoglobulin E-mediated childhood food allergy is ~8% with up to 11% of caregivers reporting food allergy symptoms. Research also suggests that 40% of children with food allergy report food allergy to multiple food allergens. Infant food allergy can result in multiple physical symptoms including colic, vomiting, reflux, bloody stool, failure to thrive, and eczema, and has been associated with a decreased quality of life in infants and their caregivers. Treatment options for infant food allergies are currently limited. In most situations, mothers must choose between continuing to breastfeed while attempting to avoid potential food allergens or ending breastfeeding and providing expensive hydrolyzed infant formula.

Breastfeeding affects mortality in children under the age of 5 years old reducing episodes of diarrhea and respiratory infections, and decreasing hospital admissions by up to 70%. The Lancet series on breastfeeding quantified the global economic health impact of breastfeeding on healthcare due to infant illness and mortality. Of the estimated 130 million live births per year globally, 820,000 infant deaths, 87% of which are under 6 months old, could be mitigated with improved breastfeeding practices. The Lancet report projects that a 10% increase in exclusive breastfeeding up to 6 months would translate to an estimated $312 million in healthcare savings in the US alone. Long-term (up to 2 years), additional breastfeeding benefits would impact treatment costs for infants and toddlers as much as $2.45 billion in the US.

Many breastfeeding women are led to believe that they should not eat certain foods (e.g., dairy) because this might lead to food intolerance in their infants. Without a method to directly test human milk, mothers will methodically cut out whole food groups (most of them extremely healthy) without realizing that the true problem is going undetected. This often starts with dairy and quickly spirals until her diet is very limited. A total elimination diet is typical for this community. Many women reduce their intake down to as few as five foods (i.e., chicken, mango, coconut oil, spinach, and potato). This extreme dietary restriction puts mothers and infants at risk for nutritional deficiencies with potential life-long effects.

Currently, there is no mechanism available for mothers to know what allergens are present in their milk. Food diaries are inadequate as dietary protein only enters breastmilk a portion of the time and is present in the milk for a variable amount of time depending on several factors including metabolism, nursing schedule and unknown individual characteristics. A simple at-home test strip would empower women to continue breastfeeding by removing the mystery of the allergens present. Mothers and pediatricians could use this information to determine what is causing reactions and then follow up to determine if informed dietary elimination made mom's milk safe. Women could then enjoy their favorite foods and be confident in feeding their infant.

Free to Feed has developed a first-in-class solution using patent-pending technology to detect food allergen proteins in human milk. With this knowledge, mothers would be able to identify the culprit and remove the food from their diets or wait for the allergen to clear from their milk prior to feeding through repeated testing. This technology hopes to empower mothers to breastfeed longer, giving both mom and baby lifelong benefits, while relieving the stress of inducing unknown effects.

Previous research has identified the presence of specific nonhuman proteins found in human milk. While an abundance of information exists on bovine proteins in human milk, very limited research exists examining the presence of soy proteins in human milk. Furthermore, there is no notable existing research validating the use of strips or other tools to detect food allergens in human milk.

The first aim of this research is to validate the use of this patent-pending technology, Freedom Strips, to detect bovine and soy-based food allergen proteins in human milk with the goal that women will be able to test their milk for common antigens (e.g., dairy) and make informed decisions as to whether the milk should be fed to their infants. This will benefit mothers and babies on a global scale as it will enable women to quickly and easily determine if their milk is safe to feed their infants. A second related aim is to add to current literature by identifying bovine- and soy-derived peptides in human milk after maternal consumption of these foods.

One hypothesis explaining the discomfort and increasingly distressed behavior of infants when consuming human milk containing food allergens relates to potential changes in the gastrointestinal microbiome. There is limited information on the relationship between maternal cow's milk and soy consumption and the gastrointestinal microbiome of mothers and their offspring. Therefore, the third aim of this study is to explore the impact of maternal cow's milk and soy consumption on breastmilk and maternal/infant gastrointestinal microbiomes.

Furthermore, elimination diets, dietary challenges and food reintroduction can put a significant amount of stress on mothers of children with infant food allergies. More research is needed examining how maternal stress levels might change throughout this process. A fourth aim of this study is to examine and compare maternal stress levels during dietary elimination and food challenge periods.

The proposed research study will build upon previous literature by increasing our knowledge related to the detection and identification of nonhuman proteins, specifically bovine and soy, in human milk. This study is unique because it will include a dietary intervention with increasing doses of soy or bovine milk examining how the amount of intake of a food allergen may impact protein detection. It also unique because it includes the investigation of maternal stress and maternal/infant GI microbiomes, both of which may provide more insight on the mechanisms and outcomes of infant food allergies. While our research lab has experience in investigating a variety of factors related to human milk and the microbiome, this study is unique from all other studies currently being done at the University of Idaho.

This study will consist of a randomized, cross-over, dietary intervention research design comprising a 5-day run-in period, two 3-day dietary interventions with a 2-day washout period between them, and a final 2-day washout period after the 2nd intervention. 40 mother-offspring dyads will be recruited to participate. Participants will be randomly assigned to order of intervention. Demographic and health data will be collected at baseline (d0) as will information related to typical infant crying patterns and maternal stress (Perceived Stress Scale). Baseline data collection will also include collection of a human milk sample (approximately 10 mL), a optional maternal stool sample, and an optional infant stool sample. Participants will complete two 24-hour dietary recalls during baseline collection (day 0) rather than one to obtain typical dairy and soy intake.

Run-in elimination period: After baseline collection, both groups will undergo a 5-day run-in period during which time half the subjects will eliminate soy and the other half will eliminate cow's milk. Participants will be provided with a list of foods and ingredients to avoid during this time facilitated by a registered dietitian. During these 5 days, participants will complete a daily compliance check and indicate any soy or bovine products/foods that they may or may not have consumed. On d5 of this run-in period, participants will again provide samples of milk and maternal and infant stool and will complete the Perceived Stress Scale.

Dietary intervention period I: After completing the run-in period, the women will consume 200 mL, 300 mL, and 400 mL of bovine milk or soy milk during d1, d2, and d3 (respectively). During each dietary intervention period, participants will provide 3 samples of milk (approximately 10 mL each) each of the 3 days (12 samples total), 1 maternal stool sample, and 1 infant stool sample. Daily logs will be kept to ascertain dairy and soy intake compliance, infant crying and fussiness, and maternal/infant stooling patterns. On the third day of the dietary intervention, mothers will again complete the Perceived Stress Scale.

Washout period I: Both dietary intervention periods will be followed by a 2-day washout period during which time participants will continue to eliminate bovine or soy containing foods and ingredients. Participants will also complete daily surveys indicating infant behavior and maternal/infant GI symptoms during this washout period.

Dietary intervention period II: After this, each subject will consume 200 mL, 300 mL, and 400 mL of bovine milk or soy milk (which ever they did not consumer in the first intervention period) during d1, d2, and d3 (respectively). Data and samples collected during intervention I will be collected during intervention II.

Washout period II: The second dietary intervention period will be followed by a 2-day washout period during which time they will continue to eliminate the food eliminated in intervention period II. Infant behavior and maternal/infant GI symptoms will again be recorded daily by participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18 years or older
* Ability to drive to Boise, Idaho or Moscow, Idaho or New York, New York
* Must be currently lactating or breastfeeding
* Mothers of infants aged 0-12 months
* Willing to provide samples of human milk
* Willing to consume 1-2 cups of soy milk and cow's milk daily for 3 days each

Exclusion Criteria:

* Individuals who are unable or unwilling to consume bovine or soy milk
* Individuals unwilling or unable to provide samples of human milk
* Individuals unable to speak and read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Soy proteins/peptides in human milk | 4 hours post intervention
  This will be measured using a proprietary test strip developed for this purpose as well as LC-MS methodology.
Soy proteins/peptides in human milk | 2 hours post intervention
  This will be measured using a proprietary test strip developed for this purpose as well as LC-MS methodologies.
Bovine proteins/peptides in human milk | 4 hours post intervention
  This will be measured using a proprietary test strip developed for this purpose and using LC-MS methodologies.
Bovine proteins/peptides in human milk | 2 hours post intervention
  This will be measured using a proprietary test strip developed for this purpose and using LC-MS methodologies.

SECONDARY OUTCOMES:
Maternal Stress | Measured at baseline (Day 0) and Days 5, 8, 15, and 18 of the 20-day study. Days 5 and 15 correspond to 5 days post dietary elimination of cow or soy and days 8 and 18 correspond to 3 days post dietary intervention with cow's milk or soy milk.
  Measurement of maternal perceived stress levels via the Perceived Stress Scale. The Perceived Stress Scale provides levels of perceived stress on a scale of 0 to 40 with higher scores indicating higher levels of perceived stress.
Human Milk Microbiome | Will be assessed on human milk samples collected at baseline (day 0), after the 5-day dietary elmination/run-in periods (days 5,/15), and on the third day of the 3-day dietary intervention periods (days 8/18).
  Measured using full length 16s rRNA gene sequencing methods.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Idaho, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share unidentified data.

REFERENCES:
- [Background] Quigley MA, Carson C. Breastfeeding in the 21st century. Lancet. 2016 May 21;387(10033):2087-2088. doi: 10.1016/S0140-6736(16)30534-7. No abstract available. PMID 27301815
- [Background] Rollins NC, Bhandari N, Hajeebhoy N, Horton S, Lutter CK, Martines JC, Piwoz EG, Richter LM, Victora CG; Lancet Breastfeeding Series Group. Why invest, and what it will take to improve breastfeeding practices? Lancet. 2016 Jan 30;387(10017):491-504. doi: 10.1016/S0140-6736(15)01044-2. PMID 26869576
- [Derived] Partridge CL, Paullin TR, Kim BJ, Dallas DC, Williams JE, McGuire MA, Kaur H, McGuire MK. Detection of bovine milk-, but likely not soy-derived, peptides in human milk after maternal consumption of bovine milk and soy beverage: a randomized, cross-over, dietary intervention trial. Front Nutr. 2025 Oct 23;12:1642177. doi: 10.3389/fnut.2025.1642177. eCollection 2025. PMID 41211220